CLINICAL TRIAL: NCT07011784
Title: Postural Stability in Older Women Following Online Dance Classes With Blood Flow Restriction
Brief Title: Dance and Blood Flow Restriction as Balance Training for Older Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Andreas Bergdahl, Associate Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30016017
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Older Adults, Balance; Dance; Blood Flow Restriction (BFR) Training Effects; Telehealth; Postural Stability; Older Adults at Risk of Falling; Older Adults (65 Years and Older); Balance Training Group; Online Physical Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dancing control (Active Comparator): The control group will complete online dance classes with the same dose, frequency and duration as the experimental group. They however will not wear blood flow restriction cuffs during the classes.
  Interventions: Other: Dance classes alone
- Dancing blood flow restriction (Experimental): Participants in the blood flow restriction group will wear elasticized bands during the online dance classes. They will put them on before warm-up and take them off before cool-down.
  Interventions: Other: Blood flow restriction in combination with dance classes; Other: Dance classes alone

INTERVENTIONS:
Other: Blood flow restriction in combination with dance classes — Blood flow restriction in combination with online ballet and modern-style dance classes to test if the balance of older women can be improved. Participants will wear 5 centimetre elasticized blood flow restriction bands on their proximal thighs throughout the online ballet-modern dance classes. Tightness levels will be set at a 7/10 of the perceived tightness scale used by Wilson et al. (2013), with a total restriction time of approximately 60 minutes, twice per week.
  Arms: Dancing blood flow restriction
Other: Dance classes alone — Online ballet and modern-dance inspired classes will be held on Zoom twice per week for 75 minutes. The sessions will span a 12 week time frame. All classes will begin with a warm-up, 1 plie exercise, 1 tendu exercise, a travelling ballet-inspired exercise, 1 travelling Graham or Limón modern dance exercise and a seated cool-down.

SUMMARY:
Falls are one of the leading causes of hospitalization and mortality among older adults (aged 65+) in Canada. Falls result from postural instability following age-related declines in muscle strength which begin in the 5th decade of life. Older women have higher rates of injury from falls due to greater deterioration of bone mass density and lower levels of physical activity when compared to men. Participation in physical activity and exercise has been shown to slow these age-related declines in postural stability by improving muscle function as well as proprioceptive and sensory systems, however the majority of older women are inactive. Dance has been used to inspire physical activity uptake among older women, and is particularly good for balance due to its both sensory and motor aspects that focus on precise execution of movement. Dance interventions have been found to improve postural stability and balance confidence.

Post-pandemic, online dance classes have provided greater accessibility to exercise interventions aimed at promoting balance. These help reach women facing transportation barriers, who have a fear of exercising with others, women with time-consuming caregiver roles at home etc. While beneficial, the intensity of online classes must be lower to ensure safety, thereby limiting physiological stimulus for adaptations. As typically higher intensity exercise is needed to promote muscle strength there may not be adequate stimulus for adaptations. Furthermore, there is little evidence of strength gains even from in-person dance classes. Blood flow restriction may offer an easy and cost-effective way to mimic higher intensity exercise and boost training benefits. Blood flow restriction has been found to boost strength during low-intensity resistance training, but there is little information on adaptations after balance training or potential transfer to reduce the risk of falls.

This 12-week online exercise intervention investigates whether blood flow restriction during dance classes can augment strength, dynamic balance and postural stability of older women aged 65 years and above. Two groups of older women will participate in twice weekly 75 minute ballet and modern-dance classes over Zoom. One group will be randomized to wear 5 centimeter elasticised blood flow restriction bands on their proximal thighs during the classes. Bands will be tightened to a 7/10 of perceived tightness.

Postural stability will be assessed using 9, 30-second trials of quiet standing on a force platform in conditions of eyes-open, eyes-closed and on a foam block - trials will be staggered to reduce fatigue effects. Trials will also be video recorded for kinematic analysis of shoulder and hip displacement using Kinovea.

Dynamic balance will be assessed using the Star Excursion Balance Test. Participants will be asked to stand on one foot in the middle of the star and reach their other leg as far as they can above the line. The distance the participant reaches in each direction will be recorded and normalized by limb length.

Strength will be assessed using the 30-second Sit-to-Stand test and Calf-Raise Senior test. Both tests involve participants doing the maximum number of repetitions possible within a 30-second time frame.

Finally scales of fears of falling and overall perceptions of health will be collected.

It is expected that this study will have great practical implications as the accessibility of this program can provide opportunities to older adults from various remote locations to increase their levels of physical activity in a safe manner. The affordability may also aid in adoption by community health and recreation centers as an easy-to-implement program that helps to reduce the risk of falls of older women, thereby promoting independence and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 65 years old
* Able to visit Concordia University for all testing sessions
* Access to a device with a webcam, Zoom and stable internet
* No contraindication for physical activity from their physician

Exclusion Criteria:

* Occurrence/onset of a stroke, vertigo, concussion or lower-extremity injury during the 12-week intervention period
* Presence of venous thromboembolism, peripheral vascular disease or sickle cell anemia

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in distance reached in each direction (from pre-mid-post) on the Star Excursion Balance Test, normalized by limb length | Comparing pre testing (week 0) to mid testing (week 6) and post-testing (week 12).
Change in number of repetitions on the Calf-Raise Senior test from pre-mid-post | Comparing pre testing (week 0) to mid testing (week 6) and post-testing (week 12).
Change in number of repetitions on a 30 second Sit-to-Stand test from pre-mid-post | Comparing pre testing (week 0) to mid testing (week 6) and post-testing (week 12).
Change postural stability during 30 second trials of quiet standing (conditions: eyes open, eyes closed, foam) | Comparing pre testing (week 0) to mid testing (week 6) and post-testing (week 12).
  Videos of the quiet standing task will also be recorded for kinematic analysis of shoulder and hip sway using markerless motion capture software.

SECONDARY OUTCOMES:
Change in scores from pre-mid-post on the Falls Efficacy Scale-International and Activities Specific Balance Confidence Scale | Comparing pre testing (week 0) to mid testing (week 6) and post-testing (week 12).
Change in scores from pre-mid-post on the Short-Form Health Survey (SF-36) | Comparing pre testing (week 0) to mid testing (week 6) and post-testing (week 12).

OTHER OUTCOMES:
Attendance rate to both live online and recorded dance classes throughout the 12-week intervention | During the 12-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No